CLINICAL TRIAL: NCT03969979
Title: Assesment of the Testicular Effects of Epididymo-orchitis in Boys Via Elastograpy
Brief Title: Elastography in Boys With Epididymo-orchitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Irem Inanc, Resident Doctor, Trakya University Pediatric Surgery Department, Trakya University
Other Study IDs: ccer epididimoorsit
Record Dates: First submitted 2019-05-25; First posted 2019-05-31 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Epididymo-orchitis
Keywords: epididymo-orchitis; shear wave elastography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- testis with epididymo-orchitis: The patients' previously inflamed testis with epididymo-orchitis
  Interventions: Diagnostic Test: Shear wave elastography
- healthy testis: The patients' non inflamed testis
  Interventions: Diagnostic Test: Shear wave elastography

INTERVENTIONS:
Diagnostic Test: Shear wave elastography — shear wave elastogrophy will be performed

SUMMARY:
The patients treated in our clinic for epididymoorchitis will be given scrotal shear wave elastography by the Department of Radiology and affected testis will be compared to non affected testis radiologically. Shear wave elastography is a method of ultrasonography, which allows the focused ultrasonographic wave to be directed to the selected tissue to produce deformation of the tissue and to obtain the numerical data on the tissue elasticity by measuring the speed of the wave when the tissue is recovered. The higher the wave velocity, the lower the elasticity of the tissue.

The data to be obtained by this method will be compared statistically.

DETAILED DESCRIPTION:
Epididymo-orchitis is an inflammatory disease of the epididymis and / or testis. The clinical picture is manifested by sudden onset testicular pain and swelling. The differential diagnosis of testicular torsion should be made in the pediatric age group. While urgent surgery is required in testicular torsion, treatment with epididymo-orchitis consists of antiinflammatory and cold application. Scrotal ultrasonography is used in the differential diagnosis and epididymo-orchitis is diagnosed in epididymis.

The scrotal ultrasound for the control after the patient's symptoms have regressed gives an idea about the course of the inflammatory process. In recent years, the introduction of elastography, which is an advanced ultrasound technique, has begun to suggest the evaluation of the elasticity of testis and epididymis in various scrotal diseases.

In epididymo-orchitis, a disease that is known with inflammation of the testicular parenchyma, a study evaluating whether there is a permanent change in the testicular parenchyma after inflammation has regressed is not yet available in the English literature. In this study, it is planned to evaluate the pediatric patients from this perspective and contribute to the literature with the results to be obtained.

ELIGIBILITY:
Inclusion Criteria:

* To be followed-up and treated in the Department of Pediatric Surgery at Trakya University due to epidididymo-orchitis. (Inpatient and / or outpatient clinic)
* 18 years old or younger
* Approval by the legal guardian

Exclusion Criteria:

* Bilateral epididymo-orchitis
* Testicular pathology other than epididymo-orchitis (undescended testis, testicular torsion)
* Scrotal surgery (due to epididymoorchitis or not)
* Older than 18 years old

Max Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The patients who had epididymo-orchitis unilaterally will be called and invited to our department for elastography. The volunteers whose legal guardians accept to be involve our study will be involved.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2019-09-20 (Actual); Primary Completion 2020-06-10 (Estimated); Study Completion 2020-06-20 (Estimated)

PRIMARY OUTCOMES:
diagnosis of post inflammation process | 3 months
  Shear wave elastography numbers will be analyzed statistically

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University Faculty of Medicine, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No